CLINICAL TRIAL: NCT05862922
Title: Comparison Effects of Lumbosacral Plexus Block and Sacral Plexus Block + Suprainguinal Fascia Iliaca Plane Block Combination on Perioperative Pain Measured With Analgesia Nociceptive Index Monitor on High-risk Patients Undergoing Hip Fracture Surgery
Brief Title: Comparison Effects of Two Regional Anesthetic Technique on Pain During High Risk Hip Fracture Surgery
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Recep Aksu, Professor Doctor, TC Erciyes University
Other Study IDs: 2022/707
Record Dates: First submitted 2023-05-03; First posted 2023-05-17 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Pain; Hip Fractures; Perioperative Analgesia
Keywords: analgesia nosiception index; lumbosacral plexus block; suprainguinal fascia iliaca plane block
MeSH Terms: conditions — Pain; Hip Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- lumbosacral plexus block group
  Interventions: Device: Analgesia Nosiception İndex Monitoring
- sacral plexus + suprainguinal fascia iliaca plane block group
  Interventions: Device: Analgesia Nosiception İndex Monitoring

INTERVENTIONS:
Device: Analgesia Nosiception İndex Monitoring — ANI is a monitor that can be measured continuously and non-invasively. It measures parasympathetic tone - based on electrocardiography - by analyzing minimal changes in heart rate that occur under anesthesia, in the early stages of awakening, and in each respiratory cycle of awake patients. At the end of the measurement, a value between 0-100 is obtained.
  Parasympathetic modulation (stress level, e.g., pain) is obtained with a minimum value of 0 and a maximum of 100. ANI values measured in the early period of recovery correlate with pain scores. When compared with hemodynamic parameters, it has been reported that the ANI response is more sensitive to nociceptive stimuli occurring in the intraoperative period.

SUMMARY:
In this study, our is to compare effect of lumbosacral plexus and sacral plexus + suprainguinal fascia iliaca plane block on perioperative pain via analgesia nociceptive index monitor on high-risk patients undergoing hip fracture surgery.

DETAILED DESCRIPTION:
The most preferred types of anesthesia in hip surgery are general anesthesia or neuraxial blocks. Both types have advantages as well as disadvantages. They may cause hemodynamic instability in geriatric and comorbid patient groups.

Peripheral nerve blocks have been associated with fewer complications both in the treatment of postoperative pain and in fragile, high-risk patients, making them an alternative to other anesthesia types.

It is important for patients to accurately measure their perioperative analgesic needs. There are many subjective methods for assessing pain. In the evaluation of analgesia level with Analgesia Nociception Index (ANI) monitorization, it is advantageous to evaluate the objective findings measuring parasympathetic system activity.

ANI is a monitor that can be measured continuously and non-invasively. It measures parasympathetic tone - based on electrocardiography - by analyzing minimal changes in heart rate that occur under anesthesia, in the early stages of awakening, and in each respiratory cycle of awake patients. At the end of the measurement, a value between 0-100 is obtained.

Parasympathetic modulation (stress level, e.g., pain) is obtained with a minimum value of 0 and a maximum of 100. ANI values measured in the early period of recovery correlate with pain scores. When compared with hemodynamic parameters, it has been reported that the ANI response is more sensitive to nociceptive stimuli occurring in the intraoperative period.

In the high-risk patient group who will undergo hip surgery in the Faculty of Medicine of Erciyes University, the pain sensation in patients will be evaluated using ANI in the perioperative period, after the peripheral nerve blocks have been applied to different anatomical areas that are routinely used.

The aim of this study is to objectively reveal the perioperative pain after peripheral block applications in the patient group with serious additional morbidities by using the ANI device. It is expected that this study will enable more effective analgesia control in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who will undergo hip surgery
* ASA group 3-4 patients
* Patients without allergies
* Patients without psychiatric disorders
* Patients without opioid dependence
* Patients without severe liver and kidney failure
* Patients without arrhythmia and beta-blocker use
* Patients without contraindications for peripheral blocks

Exclusion Criteria:

* Patients who do not accept peripheral nerve block
* Patients with failed peripheral nerve block
* Patients scheduled for bilateral hip fracture surgery
* Patients who have been operated on for hip fractures before
* Patients with arrhythmia and beta-blocker use
* Patients with contraindications for peripheral blocks
* Chronic opioid consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asa group of 3-4 patients older than 18 years of age who will undergo hip fracture surgery
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-11-26 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
effective analgesia control in patients with Analgesia Nociception Index (ANI) | postoperative 24 hour
  With Analgesia Nociception Index (ANI), it is advantageous to evaluate the objective findings measuring parasympathetic system activity. A value between 0-100 is obtained, Values between 50 and 70 indicate good analgesia control. According to studies on ANI, the patient feels pain below 50. If it is above 70, it means that more analgesia is provided. It is thought that pain control will be more effective with these objective data.
Comparison of the Effects of Two Regional Anesthesia Techniques on Pain in High-Risk Hip Fracture Surgery with analgesia nociception index | postoperative 24 hour

SECONDARY OUTCOMES:
visual analog scale and ANI consistency comparison | postoperative 24 hour
  Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm) Measurements from the starting point (left end) of the scale to the patients' marks are recorded in centimeters and are interpreted as their pain. The values can be used to track pain progression for a patient or to compare pain between patients with similar conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If requested by the authorities, IP addresses can be shared.
Supporting Information: Study Protocol
Time Frame: Data will be available within 12 months of study completion
Access Criteria: Data accept requests will be reviewed by an external independent Review Panel.Requesters will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Neuman MD, Feng R, Carson JL, Gaskins LJ, Dillane D, Sessler DI, Sieber F, Magaziner J, Marcantonio ER, Mehta S, Menio D, Ayad S, Stone T, Papp S, Schwenk ES, Elkassabany N, Marshall M, Jaffe JD, Luke C, Sharma B, Azim S, Hymes RA, Chin KJ, Sheppard R, Perlman B, Sappenfield J, Hauck E, Hoeft MA, Giska M, Ranganath Y, Tedore T, Choi S, Li J, Kwofie MK, Nader A, Sanders RD, Allen BFS, Vlassakov K, Kates S, Fleisher LA, Dattilo J, Tierney A, Stephens-Shields AJ, Ellenberg SS; REGAIN Investigators. Spinal Anesthesia or General Anesthesia for Hip Surgery in Older Adults. N Engl J Med. 2021 Nov 25;385(22):2025-2035. doi: 10.1056/NEJMoa2113514. Epub 2021 Oct 9. PMID 34623788